CLINICAL TRIAL: NCT06654141
Title: Influence of Healing Time on the Outcomes of Alveolar Ridge Preservation in Periodontally Compromised Extraction Sockets: a Randomized Controlled Trial
Brief Title: Influence of Healing Time on the Outcomes of Alveolar Ridge Preservation in Periodontally Compromised Extraction Sockets
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDC-2024-1
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-10

CONDITIONS: Tooth Loss
Keywords: ridge preservation; tooth extraction
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implant placement 3 months after tooth extraction (Experimental): Alveolar ridge preservation using xenograft (Bio-Oss Collagen®) and implant placement 3 months after tooth extraction
  Interventions: Procedure: Alveolar ridge preservation
- Implant placement 6 months after tooth extraction (Active Comparator): Alveolar ridge preservation using xenograft (Bio-Oss Collagen®) and implant placement 6 months after tooth extraction
  Interventions: Procedure: Alveolar ridge preservation

INTERVENTIONS:
Procedure: Alveolar ridge preservation — Alveolar ridge preservation using xenograft (Bio-Oss Collagen®) and implant placement at 2 different time intervals (3 and 6 months)

SUMMARY:
The goal of this clinical trial is to histologically, clinically, and radiographically evaluate the healing sequelae of periodontally compromised extraction sockets grafted with Bio-Oss Collagen® at 3 and 6 months following tooth extraction in molar sites. The main question it aims to answer is:

Does healing time influence the histologic, clinical, and radiographic outcomes following socket grafting (alveolar ridge preservation) in periodontally compromised extraction sockets.

Researchers will compare a healing time of 3 months to a healing time of 6 months (conventional healing duration) to see if a shorter duration is viable for implant placement.

Participants will:

Take a cone-beam computed tomography (CBCT) scan to prepare for the surgical procedure.

Undergo tooth extraction and the extraction socket will be grafted with Bio-Oss Collagen® and a collagen membrane Bio-Gide® will be placed to stabilize the graft material.

Return at 2 weeks for suture removal and either 3- or 6-months post-extraction for implant placement.

Return at 2 weeks post-implant placement for suture removal, 3 months for prosthesis fabrication, 4 months for final prosthesis loading, and 1 year post-loading.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* ASA (American Society of Anesthesia) status I or II
* Need for molar extraction due to periodontal disease with or without chronic endodontic involvement, complying with the presentation of periodontitis stage III/IV
* Radiographic evidence of a bone dehiscence on at least one socket wall, where the height of the horizontal (suprabony) component of the defect (alveolar bone crest - cement-enamel junction) is >50% of the corresponding root length as measured on CBCT scans prior to extraction (Ben Amara et al., 2021)
* Radiographic evidence of at least 3 mm of residual bone wall height
* Presence of at least one adjacent tooth to the extraction site
* Treatment plan must include tooth replacement with an implant-supported fixed dental prosthesis

Exclusion Criteria:

* Extraction of multiple adjacent teeth
* Acute infection associated with the tooth to be extracted or with adjacent teeth
* Current smokers (>10 cigarettes per day)
* Uncontrolled diabetes mellitus (HbA1c >7.0)
* Any active oral or systemic acute infections
* Currently receiving chemo- or radiotherapy or a history of radiotherapy in the head and neck area
* Diseases or medications that may compromise normal wound healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of vital bone via histomorphometric evaluation of bone core biopsies at 3 months | 3 months
  Percentage of vital bone
Percentage of vital bone via histomorphometric evaluation of bone core biopsies at 6 months | 6 months
  Percentage of vital bone

SECONDARY OUTCOMES:
Linear dimensional alterations of the alveolar ridge from the time of tooth extraction to the time of implant placement (3 months) | 3 months
  Clinical and radiographic (via CBCT) assessment. The buccal-lingual ridge width at the time of the extraction will be measured clinically using a periodontal probe (UNC-15) and prior to implant placement (3-months). The same measurements will be performed radiographically through the CBCTs taken prior to tooth extraction and prior to implant placement, utilizing a CBCT viewer software. The linear vertical alterations will be used utilizing the same methods, using fiduciary anatomical landmarks. Superimposition of the digital files obtained from the intra-oral scanner will be utilized to verify these changes clinically.
Linear dimensional alterations of the alveolar ridge from the time of tooth extraction to the time of implant placement (6 months) | 6 months
  Clinical and radiographic (via CBCT) assessment. The buccal-lingual ridge width at the time of the extraction will be measured clinically using a periodontal probe (UNC-15) and prior to implant placement (6-months). The same measurements will be performed radiographically through the CBCTs taken prior to tooth extraction and prior to implant placement, utilizing a CBCT viewer software. The linear vertical alterations will be used utilizing the same methods, using fiduciary anatomical landmarks. Superimposition of the digital files obtained from the intra-oral scanner will be utilized to verify these changes clinically.
Assessment of the mucosal healing of the extraction sites at 2 weeks using a wound healing index (1-3 scale rating) | 2 weeks following tooth extraction and alveolar ridge preservation
  Wound Healing Index.1-3 scale rating: 1) Uneventful Healing, 2) Normal healing with moderate soft tissue inflammation, erythema but no suppuration and 3) poor wound healing with significant signs of clinical inflammation and/or suppuration
Assessment of the mucosal healing after implant placement at 2 weeks using a wound healing index (1-3 scale rating) | 2 weeks after dental implant placement
  Wound Healing Index.1-3 scale rating: 1) Uneventful Healing, 2) Normal healing with moderate soft tissue inflammation, erythema but no suppuration and 3) poor wound healing with significant signs of clinical inflammation and/or suppuration
Patient reported outcomes (number of days of total or partially impaired activity) following tooth extraction | At the time of implant placement (3 or 6 months)
  Number of days of total or partially impaired activity
Patient reported outcomes (number of days of total or partially impaired activity) following implant placement | 4 months post implant placement
  Number of days of total or partially impaired activity
Patient reported outcomes (pain) 2 weeks following tooth extraction, using a Visual Analog Score for pain (0-100) | 2 weeks following tooth extraction and alveolar ridge preservation
  Visual Analog Score for pain (0-100, with 0 representing no pain, and 100 very severe pain, described as "worse pain imaginable").
Patient reported outcomes (pain) 3 months following tooth extraction, using a Visual Analog Score for pain (0-100) | 3 months following tooth extraction and alveolar ridge preservation
  Visual Analog Score for pain (0-100, with 0 representing no pain, and 100 very severe pain, described as "worse pain imaginable").
Patient reported outcomes (pain) 6 months following tooth extraction, using a Visual Analog Score for pain (0-100) | 6 months following tooth extraction and alveolar ridge preservation
  Visual Analog Score for pain (0-100, with 0 representing no pain, and 100 very severe pain, described as "worse pain imaginable").
Patient reported outcomes (patient satisfaction), using a Visual Analog Scale (0-100) | Up to 30 days post implant crown delivery
  Patients will be asked to rate their satisfaction in terms of function, comfort and esthetics, using a Visual Analog Scale (0-100, with 0 meaning "not at satisfied at all" and 100 corresponding to "perfectly satisfied").
Implant survival rate | 1 year post implant loading
  Percentage of implants still in the mouth
Marginal bone level changes | 1 year post implant loading
  Measured in millimeters using standardized parallel technique intraoral radiographs

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China

REFERENCES:
- [Background] Avila-Ortiz G, Elangovan S, Kramer KW, Blanchette D, Dawson DV. Effect of alveolar ridge preservation after tooth extraction: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):950-8. doi: 10.1177/0022034514541127. Epub 2014 Jun 25. PMID 24966231
- [Background] Dai A, Li HY, Kang S, Lin R, Huang JP, Mao F, Ding PH. Effect of alveolar ridge preservation at periodontally compromised molar extraction sockets: A retrospective cohort study. J Periodontol. 2025 Jan;96(1):9-20. doi: 10.1002/JPER.24-0064. Epub 2024 Jun 17. PMID 38884702
- [Background] Ben Amara H, Kim JJ, Kim HY, Lee J, Song HY, Koo KT. Is ridge preservation effective in the extraction sockets of periodontally compromised teeth? A randomized controlled trial. J Clin Periodontol. 2021 Mar;48(3):464-477. doi: 10.1111/jcpe.13412. Epub 2021 Jan 19. PMID 33316099
- [Background] Zellner JW, Allen HT, Kotsakis GA, Mealey BL. Wound healing after ridge preservation: A randomized controlled trial on short-term (4 months) versus long-term (12 months) histologic outcomes. J Periodontol. 2023 May;94(5):622-629. doi: 10.1002/JPER.22-0187. Epub 2023 Jan 10. PMID 36527199
- [Background] Couso-Queiruga E, Weber HA, Garaicoa-Pazmino C, Barwacz C, Kalleme M, Galindo-Moreno P, Avila-Ortiz G. Influence of healing time on the outcomes of alveolar ridge preservation using a collagenated bovine bone xenograft: A randomized clinical trial. J Clin Periodontol. 2023 Feb;50(2):132-146. doi: 10.1111/jcpe.13744. Epub 2022 Nov 18. PMID 36345818